CLINICAL TRIAL: NCT07006740
Title: A Multicenter, Non-Randomized Controlled Observational Study on the Safety and Effectiveness of Unilateral MR-Guided Focused Ultrasound Thalamotomy for Essential Tremor
Brief Title: Safety and Effectiveness of Unilateral MR-Guided Focused Ultrasound Thalamotomy for Essential Tremor
Acronym: BJGB-ET
Status: Not yet recruiting | Type: Observational
Sponsor: meishanshan (Other)
Collaborators: Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor-Investigator, meishanshan, Associate Chief Neurologist, Department of Neurology, Beijing Gaobo Hospital, M.D., Ph.D., Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: RP2025-023-002; BJGBYY-IIT-LCYJ-2025-023 (Other: Beijing GoBroad Hospital)
Record Dates: First submitted 2025-05-30; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; MRgFUS; Focused Ultrasound; VIM Thalamotomy; Noninvasive Neuromodulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRgFUS Group: Participants in this group will undergo unilateral MR-guided focused ultrasound (MRgFUS) thalamotomy targeting the ventral intermediate nucleus (VIM) of the thalamus. The procedure is non-invasive and performed under MRI guidance. Subjects will be followed prospectively for 12 months to assess changes in tremor severity, quality of life, and safety outcomes.
  Interventions: Procedure: MR-guided Focused Ultrasound Thalamotomy
- Medical Therapy Group: Participants in this group will receive standard medical therapy for essential tremor, which may include beta-blockers (such as propranolol), primidone, or other clinically indicated medications. Treatment plans will be determined by the attending physicians according to routine clinical practice. Participants will be followed for 12 months to assess changes in tremor severity, quality of life, and safety outcomes, consistent with the surgical treatment group.

INTERVENTIONS:
Procedure: MR-guided Focused Ultrasound Thalamotomy — This intervention involves a unilateral magnetic resonance-guided focused ultrasound (MRgFUS) thalamotomy targeting the ventral intermediate nucleus (VIM) of the thalamus. The procedure is non-invasive and uses MRI guidance to deliver focused ultrasound energy to ablate the target area. It is performed without surgical incisions or implanted devices. The intervention is intended for patients with medication-refractory essential tremor. Participants receiving this intervention will be followed for 12 months to assess efficacy and safety.
  Groups: MRgFUS Group

SUMMARY:
Essential tremor (ET) is one of the most common movement disorders, significantly impacting patients' quality of life. Many patients do not respond well to medication or cannot tolerate side effects, leaving limited treatment options. Magnetic Resonance-guided Focused Ultrasound (MRgFUS) is a noninvasive, targeted therapy that offers a promising alternative to surgical procedures such as deep brain stimulation.

This study is a multicenter, non-randomized controlled observational study designed to evaluate the safety and effectiveness of unilateral MRgFUS thalamotomy targeting the ventral intermediate nucleus (VIM) in patients with medication-refractory essential tremor. Participants will be divided into two groups based on clinical evaluation and patient preference: the treatment group receiving MRgFUS and the control group receiving standard medical therapy. Both groups will undergo regular follow-up for one year.

The primary outcome is improvement in tremor severity as measured by the Fahn-Tolosa-Marin Tremor Rating Scale and the Clinical Rating Scale for Tremor. Secondary outcomes include quality of life, cognitive and emotional status, and treatment-related adverse events.

Eligible participants are adults aged 22 years or older who have a confirmed diagnosis of essential tremor and are significantly impaired despite medication. The goal is to assess whether MRgFUS provides sustained tremor relief and improves quality of life in comparison to standard care, while maintaining an acceptable safety profile.

DETAILED DESCRIPTION:
Essential tremor (ET) is a progressive neurological disorder characterized primarily by action tremor affecting the upper limbs, head, or voice. Although ET is commonly treated with medications such as beta-blockers and anticonvulsants, a significant proportion of patients are either refractory to or intolerant of pharmacologic therapies. For these patients, surgical interventions such as deep brain stimulation (DBS) or thalamotomy may be considered. However, these procedures are invasive and associated with considerable risks and costs.

Magnetic resonance-guided focused ultrasound (MRgFUS) is a novel, non-invasive technology that enables precise thermal ablation of brain targets, such as the ventral intermediate nucleus (VIM) of the thalamus, under real-time MRI guidance. MRgFUS offers advantages such as immediate effect, no need for implants, and lower complication rates.

This multicenter, non-randomized, controlled observational study aims to evaluate the real-world effectiveness and safety of unilateral MRgFUS VIM thalamotomy in patients with medication-refractory ET. Patients will be allocated into treatment or control groups based on clinical judgment and patient preference. The study will focus on assessing improvements in tremor severity, quality of life, and treatment safety over a 12-month follow-up period. The findings will provide evidence on the utility of MRgFUS as a non-invasive therapeutic option and help inform future clinical decision-making for ET management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Diagnosis of essential tremor confirmed by clinical criteria
* Medication-refractory tremor with significant functional impairment
* Ability to provide informed consent
* Willingness to undergo follow-up assessments for 12 months

Exclusion Criteria:

* History of other neurological disorders (e.g., Parkinson's disease)
* Presence of unstable medical conditions (e.g., uncontrolled hypertension)
* Contraindications to MRI (e.g., implanted metal devices)
* Severe cognitive impairment or psychiatric illness
* Pregnancy or breastfeeding

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 22 years and older) diagnosed with medication-refractory essential tremor. Participants will be recruited from outpatient neurology clinics at multiple centers in China. All participants must be capable of providing informed consent and willing to complete a 12-month follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in Tremor Severity Assessed by the Fahn-Tolosa-Marin Tremor Rating Scale (FTM) | Baseline and 12 months
  Tremor severity will be assessed using the Fahn-Tolosa-Marin Tremor Rating Scale (FTM), which evaluates tremor at rest, with posture, and during action. The scale ranges from 0 to 144, with higher scores indicating more severe tremor.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article (after de-identification) will be shared upon reasonable request. Data will be available to qualified researchers with a data use agreement, starting 6 months after publication and for up to 3 years.
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting documents will be available beginning 6 months after publication and will be available for up to 3 years.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the de-identified individual participant data and related documents (such as the study protocol and statistical analysis plan). Data will be shared upon reasonable request under a data use agreement. Requests can be submitted by contacting the study sponsor at [your email address here].